CLINICAL TRIAL: NCT01025323
Title: Lifestyle Intervention in Multinational Hispanics With Prehypertension
Brief Title: Study of Hispanics to Assess Risk Prevention in Prehypertension
Acronym: SHARPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to difficult recruitment and retention of subjects, these were attributed by subjects to conflict with their job schedule.
Sponsor: Florida Heart Research Institute (Other)
Responsible Party: Principal Investigator, Maria Canossa Terris MD, Medical Director, Florida Heart Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FHRI 2007-02
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Pre-Hypertension
Keywords: Pre hypertension; Lifestyle modification; DASH diet
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal Intervention Group (Active Comparator): Participants in this arm receive advice and printed guidelines but no counseling or systematic instruction.
  Interventions: Behavioral: Lifestyle modification
- Enhanced Intervention Group (Active Comparator): Participants in this group receive advice and the same printed guidelines as the Minimal Intervention Group, together with dietary and physical activity counseling provided by a dietician and/or coordinator, periodic professional reviews of their progress and systematic instruction.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Behavioral: Lifestyle modification — DASH diet and exercise advice
  Other Names: MIG
  Arms: Minimal Intervention Group
Behavioral: Lifestyle modification — DASH diet, exercise with systematic instruction by a dietician and/or coordinator
  Other Names: EIG
  Arms: Enhanced Intervention Group

SUMMARY:
The purpose of this study is to assess the efficacy of lifestyle modification in reducing blood pressure values in Hispanics at risk for hypertension.

DETAILED DESCRIPTION:
In this study participants (who have prehypertension as defined as systolic blood pressure - the upper number- 130-139 mmHg and diastolic blood pressure 85-89mmHg- the lower number-) are randomly assigned to one of two groups:

the Minimal Intervention Group- participants receive advice and printed guidelines only but no counseling or personalized instruction, or the Enhanced Intervention Group- participants receive advice and the same printed guidelines as the minimal intervention group, together with dietary and physical activity counseling provided by a dietician and/or coordinator, periodic professional reviews of their progress and personalized instructions.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic men and women age 18 or older
* Mean baseline SBP 130-139 mmHg and DBP 85-89 mmHg on screening visits 1&2
* Subjects who have access to a telephone
* Subjects who have read, signed and received a copy of the informed consent form prior to the initiation of any study procedures and who agree to participate in all aspects of the study
* Subjects who are willing and capable of complying with the requirements of the study

Exclusion Criteria:

* BMI > 35
* Pregnant or breast feeding
* Currently taking any anti-hypertensive medications
* History of cardiovascular disease (Stroke, MI, PCI, CABG)
* Current symptoms of angina or peripheral vascular disease by Rose questionnaire
* Fasting glucose ≥ 126mg/dl) or a history of diabetes and use of antidiabetic medication
* Use of oral corticosteroids > 5days/month on average
* Consumption of more than 21 alcoholic drinks per week or consumption of 6 or more drinks on one occasion twice or more per week in the past 3 months prior to screening visit
* Use of weight loss medications (prescription or over the counter) in the past 3 months prior to screening visit 1 or body weight change > 15 pounds in the 3 months prior to screening visit
* Currently undergoing or planning to undergo treatment for a neoplastic disease
* Clinical significant laboratory test results that are indicative of a serious medical condition
* Renal Insufficiency (GFR<60ml/min as estimated using Cockcroft -Gault formula)
* Any orthopedic or rheumatologic problems that might limit a subject's ability to participate in the physical activity component of the intervention
* Any medical condition which in the judgment of the Investigator places the subject at risk due to his/her participation in the study, is likely to prevent the subject from complying with the requirements of the study or completing the study or which may jeopardize the evaluation of efficacy or safety
* Planning to leave area prior to the anticipated end of participation
* Current participation in another research study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To test the effect on systolic blood pressure on the Enhanced Intervention Group compared to the Minimal Intervention Group | 6 months

SECONDARY OUTCOMES:
The test the effect on systolic and diastolic blood pressure,lipid profile, glucose level, c-reactive protein and body mass index of the Enhanced Intervention Group in comparison to the Minimal Intervention Group | 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Canossa-Terris, MD, Principal Investigator — Florida Heart Research Institute
Locations (1):
- Florida Heart Research Institute, Miami, Florida, United States